CLINICAL TRIAL: NCT01886313
Title: A DOUBLE BLIND, RANDOMIZED, VEHICLE-CONTROLLED, PARALLEL-GROUP EVALUATION OF CIVAMIDE (ZUCAPSAICIN) 0.01% AND VEHICLE NASAL SPRAYS IN THE TREATMENT OF POSTHERPETIC NEURALGIA OF THE TRIGEMINAL NERVE
Brief Title: Civamide Nasal Solution for Postherpetic Neuralgia of the Trigeminal Nerve
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WL-1001-07-01
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Postherpetic Neuralgia
Keywords: Herpes Zoster; Postherpetic Neuralgia; Shingles; Civamide; Zucapsaicin; Neuropeptides; TRPV-1
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Civamide Nasal Spray (Active Comparator): Civamide Nasal Spray 0.01% 20ug/dose (20ul), 10ul in each nostril, twice daily, for 6 weeks
  Interventions: Drug: Civamide Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): Placebo Nasal Spray 10ul in each nostril, twice daily, for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Civamide Nasal Spray
  Arms: Civamide Nasal Spray
Drug: Placebo
  Arms: Placebo Nasal Spray

SUMMARY:
Herpes zoster (commonly referred to as "shingles") results from the reactivation of the varicella-zoster virus acquired during a primary infection, usually chickenpox. The virus lays dormant in the cells of the nerves until activated. Once activated, patients develop a characteristic red blistering rash which crusts and heals in 2 - 4 weeks. Postherpetic neuralgia (PHN), the term for pain persisting after the herpes zoster (HZ) eruption heals, is the most common and most feared complication of herpes zoster infection. The drug, Civamide is thought to desensitize the nerves and decrease the pain of PHN. This is the pharmacologic rationale for its use in the nose in postherpetic neuralgia of the trigeminal nerve, a nerve that is in the nose and transmits pain from the face. The objective of this study is to evaluate the safety and efficacy of intranasally administered Civamide (0.01%) for the treatment of moderate to severe daily pain associated with postherpetic neuralgia of the trigeminal nerve. Neuropathic pain must have persisted for ≥ 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the screening procedures.
2. Subject is in generally good health other than a history of postherpetic neuralgia, determined by pre-study medical evaluation (medical history, physical examination including examination of the treatment area, and vital signs) and without evidence of underlying unstable acute or chronic systemic disease, e.g. diabetes.
3. Subject has experienced on average, moderate to severe chronic postherpetic neuralgia restricted to the distribution of the affected trigeminal nerve or its divisions for at least 12 months after healing of a herpes zoster skin rash.
4. Subject has Average Daily Pain Score of 4 or higher on the 11-point numeric rating scale during the 7-Day Baseline Period.
5. Males or females between 21 to 80 years of age, inclusive.
6. Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (abstinence, hormonal contraceptives, diaphragm with spermicide, condom with spermicide, or intrauterine device) throughout the study or females of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year). A negative urine pregnancy test must be confirmed at screening for all female subjects who are not surgically sterile.
7. The subject agrees not to begin any new concomitant medications during their participation in study.

Exclusion Criteria:

1. Subject has a history of frequent headache or other painful conditions, other than that associated with PHN, within the past 30 days that has required or is expected to require the additional use (beyond stable daily doses) of prescription or over the counter pain relief medication, such as non-steroidal anti-inflammatory agents, including COX-2 inhibitors, systemic opiates or derivatives, or acetaminophen more than 2 times per week during the study. Concurrent medications and stable dose requirements are listed in Table 3.
2. Clinical, historical or previous laboratory evidence of significant cardiovascular, renal, gastrointestinal, pulmonary, hepatic, endocrine, neurological, psychological, or other systemic disease that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk to the subject.
3. Presence of a significant nasal disorder.
4. Subject is immunocompromised (e.g. AIDS, significant oncologic disease, immunocompromising medications, etc.).
5. Subject received neurolytic or neurosurgical therapy for this or previous episodes of postherpetic neuralgia.
6. Use of any restricted medication within the given time period prior to the Baseline Period and throughout the study (see Table 1).
7. Subject has a history of alcohol and/or drug abuse within the past year.
8. Subject has previously participated in a Civamide study.
9. Subject has participated in another investigational study or taken another investigational drug within the past 30 days.
10. Subject has difficulty distinguishing his/her PHN head pain from other types of head pain, such as tension-type headaches.
11. Known hypersensitivity to or contraindication to the use of Civamide (zucapsaicin), capsaicin (Zuacta®, Zostrix®, Zostrix-HP®, Axsain®, or related products) or to any excipient of the clinical formulation.
12. Initiation of a medication, discontinuation of a medication or change in regimen of existing medication(s) or therapies less than the required period of stable dosing prior to entering the Baseline Period. (See table 2.)
13. If, for any other reason, the subject is not deemed to be suitable by the Investigator, they should not be enrolled.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - California Medical Clinic for Headache, Santa Monica, California
  - Sun Rise Medical, Lauderdale Lakes, Florida
  - Meridien Research, Tampa, Florida
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Furture Search Trials of Neurology, LP, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 5 centers in the United States.
Pre-assignment Details: Subjects who met a minimum average daily pain score of ≥4 were equally randomized into either active or placebo groups.
Groups:
- Double Blind Treatment Period Civamide Nasal Spray: Civamide Nasal Spray 0.01% 20ug/dose (20ul), 10ul in each nostril, twice daily, for 6 weeks
  Civamide Nasal Spray
- Double Blind Treatment Period Placebo Nasal Spray: Placebo Nasal Spray 10ul in each nostril, twice daily, for 6 weeks
  Placebo
Period: Overall Study
Arm/Group | Double Blind Treatment Period Civamide Nasal Spray | Double Blind Treatment Period Placebo Nasal Spray
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind Treatment Period Civamide Nasal Spray | Double Blind Treatment Period Placebo Nasal Spray | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 5 | 2 | 7
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Pain Score
Description: The change in the Average Daily Pain Score (11-point Numeric Rating Scale (NRS)) from the Baseline Period to the Average Daily Pain Score of the last week of the Treatment Period. The minimum score is 0 and the maximum score is 10. A score of 0 indicates no pain while a score of 10 indicates worst possible pain.
Time Frame: 6 weeks
Population: 1 patient withdrew early from study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind Treatment Period Civamide Nasal Spray | Double Blind Treatment Period Placebo Nasal Spray
Number analyzed (Participants) | 6 | 5
units on a scale
  Baseline | 6.4 (0.84) | 5.2 (1.02)
  Week 6: number analyzed (Participants) | 5 | 5
  Week 6 | 5.3 (1.24) | 3.1 (2.13)

ADVERSE EVENTS:
Time Frame: 6 week Treatment Period, 2 week Post Treatment Observation Period
Arm/Group | Double Blind Treatment Period Civamide Nasal Spray | Double Blind Treatment Period Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Treatment Period Civamide Nasal Spray (N=6) | Double Blind Treatment Period Placebo Nasal Spray (N=5)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject was hospitalized
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Treatment Period Civamide Nasal Spray (N=6) | Double Blind Treatment Period Placebo Nasal Spray (N=5)
Application Site Burning (General disorders) | 3 (11) | 1 (1)
Application Site Irritation (General disorders) | 3 (17) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0)
Eye Irriation (Eye disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No